CLINICAL TRIAL: NCT00005765
Title: Behavioral Economics of Human Drug Self-Administration
Status: Completed | Type: Observational
Sponsor: National Center for Research Resources (NCRR) (NIH)
Other Study IDs: NCRR-M01RR00109-0747; M01RR000109 (NIH)
Record Dates: First submitted 2000-06-01; First posted 2000-06-02 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2003-12

CONDITIONS: Drug Dependence
MeSH Terms: conditions — Substance-Related Disorders | interventions — Nicotine; Ethanol

STUDY DESIGN:
Observational Model: Natural History | Time Perspective: Cross-Sectional

INTERVENTIONS:
Drug: nicotine
Drug: alcohol

SUMMARY:
The objective of this protocol is to examine the utility of behavioral economics for understanding reinforcer interactions as they pertain to drug self-administration. In a series of 6 experiments, the researchers will attempt to quantify the effects of qualitatively different reinforcers (money, cigarettes, alcohol, nicotine gum) and their interactions. This work represents a continuation of research by this investigator in the area of addiction and pharmacology.

ELIGIBILITY:
Inclusion Criteria:

* Use of 20 or more cigarettes per day
* CO levels >15 ppm
* More than 12 alcohol drinks per week and beer as preferred alcoholic beverage

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult

CONTACTS AND LOCATIONS:
Locations (1):
- University of Vermont, Burlington, Vermont, United States